CLINICAL TRIAL: NCT03068260
Title: Ultrasound-guided Transmuscular Quadratus Lumborum Block for Elective Caesarean Section. A Double Blind, Randomized, Placebo Controlled Trial.
Brief Title: Ultrasound-guided Transmuscular Quadratus Lumborum Block for Elective Caesarean Section.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZUH-TQL-ECS
Record Dates: First submitted 2017-02-14; First posted 2017-03-01 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Pain
Keywords: caesarean section; postoperative pain; transmuscular quadratus lumborum block; reduction of opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride; Acetaminophen; Ibuprofen; Tablets; Morphine; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Active bilateral ultrasound-guided transmuscular quadratus lumborum (TQL) block. 60 ml ropivacaine 0,375% single shot.
  In both arms, the participants receive 1g Acetaminophen and 400 mg Ibuprofen / 100 mg Celebra. Morphine will be administered IV as part of a PCA-pump regimen or additionally after contact with the nursing staff as it is the standard treatment.
  Interventions: Drug: Ropivacaine; Drug: Acetaminophen; Drug: Ibuprofen 400Mg Tablet / Celebra 100 Mg tablet; Device: ultrasound-guided nerve block; Drug: Morphine; Device: Patient-controlled analgesia
- Placebo (Placebo Comparator): Placebo bilateral ultrasound-guided transmuscular quadratus lumborum (TQL) block. 60 ml saline single shot.
  In both arms, the participants receive 1g Acetaminophen and 400 mg Ibuprofen / 100 mg Celebra. Morphine will be administered IV as part of a PCA-pump regimen or additionally after contact with the nursing staff as it is the standard treatment.
  Interventions: Drug: Saline; Drug: Acetaminophen; Drug: Ibuprofen 400Mg Tablet / Celebra 100 Mg tablet; Device: ultrasound-guided nerve block; Drug: Morphine; Device: Patient-controlled analgesia

INTERVENTIONS:
Drug: Ropivacaine — 30 ml ropivacaine 0,375% administered on each side as bilateral TQL blocks
  Arms: Active
Drug: Saline — 30 ml saline 0,375% administered on each side as bilateral TQL blocks
  Arms: Placebo
Drug: Acetaminophen — 1 g orally administered postoperatively
Drug: Ibuprofen 400Mg Tablet / Celebra 100 Mg tablet — orally administered postoperatively
Device: ultrasound-guided nerve block — Transmuscular quadratus lumborum block, ultrasound-guided
Drug: Morphine — intravenously administered morphine via PCA-pump
Device: Patient-controlled analgesia — PCA-pump with IV-Morphine. 5 mg administered per bolus. Lock-out time and max. dosage standardized.

SUMMARY:
ECS is a very common procedure. A 1-year retrospective survey revealed a vast opioid consumption among the new mothers of approximately (mean±SD) 35±25 mg of oral morphine in the first 24 postoperative hours despite a multimodal analgesic regimen. The adverse effects of morphine are well known and include postoperative nausea and vomiting (PONV), itching, fatigue, constipation, confusion, respiratory depression and delayed mobilization. These adverse effects are unsound for the new mothers as well as the breast-fed, newborn children. This study aims to evaluate the efficacy of bilateral Transmuscular Quadratus Lumborum (TQL) block in reducing postoperative morphine consumption and pain.

DETAILED DESCRIPTION:
Every year two hundred and twenty patients undergo elective caesarean section (CS) at the department of obstetric and gynaecologic surgery at Zealand University Hospital. The vast majority of these patients undergo the surgical procedure under spinal (subarachnoid) anaesthesia with Bupivacaine with the additive Sufentanil.

There are many ways to perform a caesarean section. The techniques can vary, regarding the type of skin incision, how the abdominal wall is dissected, how the uterine incision is made, and finally in which layers are closed after the procedure.

Two common transverse skin incisions are the Pfannenstiels incision and the Joel-Cohen incision. The Pfannenstiels incision is made 2 to 3 cm cephalad to the pubic bone, slightly curved so the midportion of the incision is within the shaved area of the pubic hair. The Joel-Cohen incision is placed 3 cm caudad to the anterior intercristal line; i.e. slightly more cephalad than the Pfannenstiels incision.

If the Pfannenstiels incision is utilized, the subcutaneous layer, fascia and the parietal peritoneum are usually dissected sharply, whereas with the Joel-Cohen incision, the subcutaneous layer is only incised medially, followed by a manual separation of the lateral tissue. The fascia and peritoneum are dissected bluntly.

At Zealand University Hospital, the skin incision used for elective caesarean sections is the Joel-Cohen incision. A straight, transverse, 12 cm long incision is made through the cutaneous layer as described above. The subcutaneous layer is incised only in the most medial area, through which two small incisions are made on each side of the midline of the fascia. These incisions in the fascia are then extended laterally with a scissor. The linea alba and parietal peritoneum are opened bluntly with the fingers. Finally, all the layers of the abdominal wall are pulled apart at the angles of the incisions, opening the incision laterally.

The sensory nerve supply to the abdominal wall below the umbilicus consists of the anterior cutaneous rami of the 11th intercostal nerve, the subcostal nerve (T12), the iliohypogastric nerve (T12, L1) and the ilioinguinal nerve (L1).

From the intercostal space, the 11th intercostal nerve runs behind the costal cartilage and enters into the neurovascular plane between the internal oblique- and the transverse abdominis muscles. Just lateral to the rectus abdominis muscle, the nerve perforates the dorsal sheath of the rectus muscle and continues through the rectus muscle to end as an anterior cutaneous branch of the abdominal wall just below the umbilicus. The subcostal nerve passes under the lateral arcuate ligament, runs in front of the quadratus lumborum muscle and then perforates the transverse abdominis muscle to enter the neurovascular plane. Here the subcostal nerve divides into an anterior and a lateral branch, where the anterior branch innervates the skin in the hypogastrium. The iliohypogastric nerve emerges from the lateral border of the psoas major muscle and runs in front of the quadratus lumborum muscle behind the kidney. The nerve perforates the transverse abdominis muscle near the iliac crest and enters into the neurovascular plane between the transverse abdominis and internal oblique muscle where it divides into a lateral and an anterior cutaneous branch. The lateral branch innervates the skin of the gluteal region, whereas the anterior branch perforates the internal oblique muscle, runs between the internal and external oblique muscle until it perforates the external oblique muscle 2-3 cm cranial to the subcutaneous inguinal ring and ends as an anterior cutaneous branch to the skin of the hypogastric region. The ilioinguinal nerve initially follows the iliohypogastric nerve, just caudad to it, and sometimes communicating with it in a common nerve. After perforating the internal oblique muscle, it runs through the superficial inguinal ring and innervates the skin over mons pubis, labia majora and the upper and medial part of the thigh.

The parietal peritoneum lines the abdominal cavity and is innervated by the same spinal nerves as its corresponding region of the abdominal wall.

When entry to the abdominal cavity is achieved, an incision in the peritoneum covering the bladder is made. A superficial, transverse incision is made in the midline of the lower uterine segment. The rest of the muscular layers are dissected bluntly with a pean until entering the uterine cavity where after the incision is expanded laterally by pulling in cephalocaudal direction. The infant is delivered and placenta removed.

The visceral peritoneum covers the uterus anteriorly and posteriorly. Like the parietal peritoneum, it receives the same afferent nerve innervation as the organ it covers. On each side of the uterus, the two peritoneal sheets meet and comprise the broad ligament. The fallopian tubes run between the two sheets in the free edge of this ligament, where the peritoneum folds. On each side of the fallopian tubes, the round ligament of the uterus and the ovarian ligament arise anteriorly and posteriorly, respectively. Other ligaments that support the uterus are the cardinal ligament that attaches the cervix to the lateral pelvic wall, and the uterosacral ligament that extends backwards from the cervix to the front of the sacrum. The ovaries are held in place by the ovarian ligament (to the uterus), the suspensory ligament of the ovary (to the pelvic wall) and the mesovarium (to the broad ligament).

Like most other viscera, the uterus is innervated by sympathetic and parasympathetic fibers, as well as sensory nerve fibers. It is innervated by the uterovaginal plexus, which fibers originate from the inferior hypogastric plexus. The inferior hypogastric plexus is paired, with each half on each side of the rectum, cervix and the bladder and consists of sympathetic as well as parasympathetic fibers. Pain from the body of the uterus is considered to run with the sympathetic nerves. Afferent nerves supplying the uterus arise from T10 - T12 and L1.

The fallopian tubes are also innervated by the uterovaginal plexus, as well as the ovarian plexus. The ovaries have their afferent supply from the 10th intercostal nerve.

After fetal and placental extraction, the uterotomy is closed. Where possible, it is recommended to close the uterus in-situ. The uterus is closed with a single-layer, continuous closure. Marcain is sometimes administered subfascially where after the fascia is closed with a continuous suture. Finally, the skin is closed with an intracutaneous suture.

In the post-anaesthesia care unit (PACU) the patients are administered the multimodal analgesia regimen currently consisting of oral Acetaminophen 1g, Ibuprofen 400 mg. and Morphine 10 mg. The addition of oral Morphine 10 mg is not an international standard but has been so far agreed on locally.

The investigator's research group at Zealand University Hospital has conducted a thorough retrospective one-year survey for this patient group in order to define the quantity of the research problem. The electronic anaesthesia files, PACU files and ward files were meticulously reviewed. The survey revealed accumulated morphine consumptions in the first 24 postoperative hours of 35.7±25.0 mg of oral morphine equivalents in CS patients. This dosage should be evaluated in relation to the standardised multimodal regimen described above.

Anaesthesiologists have primarily used either epidural catheters or long-lasting opioids as the basis for the postoperative pain management of expected or manifest moderate to severe pain. An epidural blockade can be contraindicated for some patients, and might cause bladder paralysis, lower extremity paralysis, hypotension etc. Also, the epidural technique is labour-intensive in application as well as in its requirements for monitoring. Thus, the continuous epidural blockade is not a possibility of interest to the gynecologists and obstetricians at our hospital. Therefore, until recently opioids have been the sole treatment of pain, when over-the-counter medicine does not suffice. This presents a problem for the patients due to the well-known adverse effects of morphine including postoperative nausea and vomiting (PONV), itching, fatigue, constipation, confusion, respiratory depression and delayed mobilisation. These adverse effects are bad for the new mothers as well as the breast-fed, newborn children. All of these adverse effects are well known, and internationally several anaesthesia associations (ESA, ASA, ESRA, ASRA) are searching for viable alternatives that can be implemented in the daily clinical practice - alternatives with the primary focus on the wellbeing of the patient striving to ensure effective pain relief with minimal adverse effects.

In summary, there could be many potentially positive benefits related to the treatment with advanced pain-reducing techniques. Postoperative complications to surgery are more frequent in patients experiencing postoperative pain, and besides reducing the immediate postoperative pain perception, we consider reduction of the total morphine consumption and the potential of reducing development of chronic pain through better treatment of the acute pain, as very interesting and promising for the patients in our study.

To avoid or reduce postoperative pain after CS, numerous regional anaesthetic techniques have been tried. In the UK, and elsewhere, the combined spinal epidural (CSE) is used, but because of high demands of time and technical skills, and it's lack of potential to have the epidural tested with the spinal on top, this technique has never gained ground in Denmark. The ultrasound-guided (USG) or 'blind' transversus abdominis plane (TAP) block has been investigated in several studies, but with varying results. Thus, this technique has not been considered for implementation into the standard anaesthesia regimen for CS at Zealand University Hospital. In a placebo controlled trial in 2015 with patients undergoing CS, Blanco et al. found significantly lower postoperative opioid consumption and lower pain scores in the active group treated with Dr. Blanco's version of an ultrasound-guided (USG) quadratus lumborum (QL) block - named QLB which much resembles an USG version of the original blind and landmarked based TAP block. However, the exact mechanism by which Dr. Blanco's QLB block works is still not clear. The investigators now have the technical capability to improve perioperative pain management by taking advantage of USG peripheral nerve blocks (PNBs). At Zealand hospital we have concomminantly with Dr. Blanco described another so-called QL block technique. We call this technique the transmuscular QL (TQL) block. The mechanism by which the TQL block works has just been proven in a major cadaveric study. (submitted for publication Anesth Analg) USG PNBs are applied using a technique based on a thorough anatomical knowledge and real-time ultrasound images that have evolved rapidly during the last 10 years. At the Department of Anaesthesiology, Zealand University Hospital, our research group is among the leaders in Scandinavia within this specific field of interest. We want to make the use of this pain treatment technique in everyday practice wherever it is clinically indicated. The research group is headed by associate professor Jens Børglum, PhD, and he has been deeply involved in this development since 2007.

In relation to abdominal surgery, Jens Børglum and his previous research group have been involved in research that has described and evaluated the effectiveness of USG bilateral dual transversus abdominis plane (BD-TAP) blocks, USG ilioinguinal / iliohypogastric nerve blocks and, more recently, the USG TQL blocks.

Three articles concerning specifically the USG TQL block and its' application has recently been published from our group alone, showing the increasing interest and focus on the development of this particular block and the potential abilities with the future knowledge of the block.

At the Zealand University Hospital several research projects regarding the seemingly very promising analgesic efficacy of the USG TQL blockade are planned and already in the making. The Department of Anaesthesiology already conduct a PhD-study in cooperation with the Department of Urology concerning the TQL block and the management of pain in patients operated for kidney cancer (nephrectomy) and large pelvis stones (Percutaneous Nephrolithotomy, PNL). The USG TQL block has shown convincing results in a small pilot-study, concerning the above-mentioned patients with surgery in the retroperitoneal space, resulting in very low pain scores and a period without the need for opioids in up to 24 hours postoperatively.

In our other pilot-studies, the USG TQL block has shown an excellent pain-relieving effect administered as a bilateral rescue block; i.e. postoperatively after laparoscopic hysterectomy and other gynaecologic procedures as well as CS.

The TQL block is applied with the patient in the lateral position, with the flank of the side to be blocked turning upwards. The ultrasound transducer is placed in the transverse position at the posterior axillary line, just above the iliac crest, and adjusted to visualise the QL and psoas major (PM) muscles and the transverse process of vertebrae L3 or L4. The needle is subsequently inserted at the posterolateral end of the transducer and advanced in plane. The needle is then advanced through the QL muscle until the tip of the needle penetrates the investing fascia of the QL muscle. The local anaesthetic is then injected in the interfascial plane, but posterior/superficial to the transversalis fascia (TF) and between the QL and PM muscles. Confirmation of correct application can subsequently be visualized when the two muscles are seen to spread apart on the ultrasound image. The TF, which cover the antero-medial surface of the QL and the antero-lateral surface of the PM, splits in two layers at the level of the diaphragm. One layer is continuous with the inferior diaphragmatic fascia and the other continues behind the arcuate ligaments of the diaphragm to be the endothoracic fascia. This is why the lumbar application of local anaesthetic can facilitate a block of nerves within the thoracic cage. The injectate will now be in close proximity with the ventral rami of the segmental nerves in the thoracic paravertebral space and the sympathetic trunk.

As previously mentioned we have yet unpublished data from a cadaveric study in Innsbruck, December 2015, conducted by our own group. The results show a very favourable spread of injectate with the TQL block. Not only does the injected dye in this study spread to colour the ventral rami of the thoracic spinal nerves up to T9 in the thoracic paravertebral space; the injectate also spread to colour the thoracic sympathetic trunk. The visceral pain arising from the intraperitoneal organs travel via different nerves to join exactly in the thoracic sympathetic trunk before entering the central nervous system. Thus, this seem to indicate that the TQL block can be used to treat not only the pain from the incisions and tears superficially to the uterus, but also the pain from the uterus itself, and the adjacent intraperitoneal organs and structures, which is affected in patients undergoing CS. The cadaveric study has also shown that the lumbar sympathetic trunk and lumbar plexus were not affected by the injected dye. These results seem to imply that there would be minimal or no affection of ambulation or lumbar sympathectomy; i.e. no hypotension or dysfunctional bladder as can often be observed with the epidural technique. Both findings that coincides with our clinical experiences from our pilot studies.

The investigators want to perform evidence-based research using the USG TQL for patients undergoing elective CS. Our hypothesis is that the USG TQL block administered bilaterally and applied postoperatively in the PACU for the CS patients (with the spinal anaesthesia still manifest) can reduce the postoperative morphine consumption by 50 % during the first 24 postoperative hours. It is considered a block with very little discomfort for the patient, when not already anaesthetized, but even more so, when the patient is still anaesthetised in our area of interest, or at least still somewhat desensitised from the spinal anaesthesia.

All patients scheduled for a CS will be screened according to the inclusion and exclusion criteria. The suitable candidates will be asked prior to surgery, whether they want to participate in the trial. If so, following elective CS surgery, the patient will receive the block, allocated in a randomised fashion to either active LA or placebo. The block will be performed under standard postoperative monitoring by a trained and skilled physician from the department of anaesthesia. The active treatment will be a bilateral TQL block with 30 mL Ropivacaine 0.375% on each side, whereas the placebo group will receive the same volume of Saline, applied in the exact same way. The patients will all receive the same post-surgical analgesia regimen, consisting of 1 g Acetaminophen, 400 mg Ibuprofen / 100 mg Celebra, the latter with larger blood loss evaluated by the anaesthetist and obstetrician, and an IV Morphine Patient-Controlled Analgesia (PCA) - pump. In order to keep the pooled administration of local anaesthetic below the accepted maximum recommended dosage, local anaesthetic infiltration will not be performed by the surgeon. In reference to opioid consumption, it has been part of a local instruction to receive 10 mg Morphine in the PACU upon arrival here post-surgically. This is also withdrawn concerning the patients enrolled in this study, but instead the patient herself will manage the opioid treatment by activation of the PCA pump.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled for elective Caesarean Section in spinal anaesthesia.
* Have received thorough information, orally and in written, and signed the "Informed Consent" form on participation in the trial

Exclusion Criteria:

* Inability to cooperate
* Inability to speak and understand Danish
* Allergy to local anaesthetics or opioids
* Daily intake of opioids
* Local infection at the site of injection or systemic infection
* Difficulty visualisation of muscular and fascial structures in ultrasound visualisation necessary to the block administration

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women scheduled for elective caesarean section are eligible.
Enrollment: 72 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Twenty-four hours postoperatively
  Data from PCA pump and patient medical record

SECONDARY OUTCOMES:
Pain intensity (NRS 0-10/10) | At 6, 12, 24, 36, 48 hours postoperatively.
  NRS score will be recorded electronically on all morphine administrations, since all patients must enter their NRS score on the PCA pump display prior to administration of the PCA boluses.
Total morphine consumption. | At 6, 12, 36 and 48 postoperative hours.
  Data from PCA pump and patient medical record
Duration of block | Time to first opioid within the first 24 postoperative hours.
  How long time does the TQL block work
Patient satisfaction with application of the block. Satisfaction measured on NRS. | Immediately after application
  0=Complete satisfaction 10=Unmanageable dissatisfaction
The degree of morphine-related side effects. Nausea or PONV registered on CRF if any. | 48 hours
  PONV. 0-3; 0=No nausea. 3=Unmanageable nausea
Time from operation to ambulation | Within the first 24 postoperative hours
  When does the new mother ambulate. I.e. Unassisted visit at the bathroom.

CONTACTS AND LOCATIONS:
Locations (1):
- ZUH, Roskilde, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No